CLINICAL TRIAL: NCT04097678
Title: Intraoperative Radiographic Detection of Retained Surgical Sponges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Twin Cities Spine Center (Other)
Collaborators: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1290533
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-10

CONDITIONS: Surgical Sponge, Retained
Keywords: lumbar spine surgery; radiographic imaging
MeSH Terms: conditions — Foreign Bodies

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized study with two cohorts: one experimental and one control.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a semi-blinded trial. Investigators performing the surgery will know whether or not a sponge is present but the investigators reviewing the images will not. Subjects will not be told which study group they are in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retained Sponge Group (Experimental): Just prior to imaging, the surgeon will purposely place a sponge in the wound. Two radiographs will be taken of the spine (AP and Lateral views).
  Interventions: Other: Retained Surgical Sponge
- No Retained Sponge Group (No Intervention): No sponge will be placed in the wound. Two radiographs will be taken of the spine (AP and Lateral views).

INTERVENTIONS:
Other: Retained Surgical Sponge — A surgical sponge will be intentionally placed in the surgical field prior to final imaging and then removed. Postoperatively, images will be assessed for the presence or absence of a retained surgical sponge.
  Arms: Retained Sponge Group

SUMMARY:
This prospective study will determine the efficacy of intraoperative x-ray to identify retained surgical sponges. The recommended practice for finding a retained sponge is by radiography. The purpose is to find out how useful plain x-rays are in open posterior lumbar spine surgery, information which is presently unavailable. The specific aim is to compare the sensitivity (seeing a sponge when one is actually present) and specificity (not seeing a sponge when one is not present) of radiography of the surgical field for three conditions: viewing one lateral radiograph versus viewing one anteroposterior radiograph versus viewing two radiographs together, one lateral and one anteroposterior.

DETAILED DESCRIPTION:
This is a prospective, randomized study with two cohorts: one experimental and one control. Anteroposterior (AP) and lateral (LAT) radiographs are routinely obtained as standard of care during spine surgery to confirm proper implant placement. These images will be used in this study. In one-half of the study subjects, after all sponges are removed, a surgical sponge will be intentionally placed in the surgical field prior to imaging. Postoperatively, each subject's images will be assessed for the presence or absence of a retained surgical sponge. Images will be independently read by two investigators. When there is discordance, the images will be adjudicated by a third. Interobserver agreement will be quantified using the Kappa statistic. Those reading images will not have participated in the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open posterior instrumented lumbar spine surgery.
* Read and understand English.

Exclusion Criteria:

* Pregnancy.
* Patients who do not consent to research.
* Patients less than 18 years old at the time of consent.
* Do not read and understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Mehbod, MD, Principal Investigator — Twin Cities Spine Center
Locations (1):
- Twin Cities Spine Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Cima RR, Kollengode A, Garnatz J, Storsveen A, Weisbrod C, Deschamps C. Incidence and characteristics of potential and actual retained foreign object events in surgical patients. J Am Coll Surg. 2008 Jul;207(1):80-7. doi: 10.1016/j.jamcollsurg.2007.12.047. Epub 2008 May 23. PMID 18589366
- [Background] Lincourt AE, Harrell A, Cristiano J, Sechrist C, Kercher K, Heniford BT. Retained foreign bodies after surgery. J Surg Res. 2007 Apr;138(2):170-4. doi: 10.1016/j.jss.2006.08.001. Epub 2007 Feb 1. PMID 17275034
- [Background] Turgut M, Akhaddar A, Turgut AT. Retention of Nonabsorbable Hemostatic Materials (Retained Surgical Sponge, Gossypiboma, Textiloma, Gauzoma, Muslinoma) After Spinal Surgery: A Systematic Review of Cases Reported During the Last Half-Century. World Neurosurg. 2018 Aug;116:255-267. doi: 10.1016/j.wneu.2018.05.119. Epub 2018 May 26. PMID 29807184
- [Background] Viera AJ, Garrett JM. Understanding interobserver agreement: the kappa statistic. Fam Med. 2005 May;37(5):360-3. PMID 15883903
- [Background] Revesz G, Siddiqi TS, Buchheit WA, Bonitatibus M. Detection of retained surgical sponges. Radiology. 1983 Nov;149(2):411-3. doi: 10.1148/radiology.149.2.6622683.
- [Background] Jones SR, Carley S, Harrison M. An introduction to power and sample size estimation. Emerg Med J. 2003 Sep;20(5):453-8. doi: 10.1136/emj.20.5.453. PMID 12954688
- [Background] Hellbach K, Beller E, Schindler A, Schoeppe F, Hesse N, Baumann A, Schinner R, Auweter S, Hauke C, Radicke M, Meinel FG. Improved Detection of Foreign Bodies on Radiographs Using X-ray Dark-Field and Phase-Contrast Imaging. Invest Radiol. 2018 Jun;53(6):352-356. doi: 10.1097/RLI.0000000000000450. PMID 29420322

RESULTS

PARTICIPANT FLOW:
Groups:
- Retained Sponge Group: A surgical sponge will be intentionally placed in the surgical field prior to final imaging and then removed. Postoperatively, images will be assessed for the presence or absence of a retained surgical sponge.
Period: Overall Study
Arm/Group | Retained Sponge Group | No Retained Sponge Group
Started | 73 | 73
Completed | 56 | 55
Not Completed | 17 | 18
Not completed — No Radiographs Obtained During Surgery | 17 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retained Sponge Group | No Retained Sponge Group | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.2) | 63.4 (11.3) | 63.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 32 | 29 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Median (Full Range); unit: kg/m^2] | 30.4 [19.5 to 46.0] | 29.4 [17.8 to 53.7] | 30.0 [17.8 to 53.7]

OUTCOME MEASURES:

1. Primary Outcome: Accuracy
Description: Reviewer accuracy is the agreement (Cohen's Kappa) between the true condition and the readers' interpretation with 1) one lateral (LAT) image, 2) one anteroposterior (AP) image, and 3) AP and LAT images together.
Time Frame: Intraoperative
Measure: Number; unit: Cohen's Kappa
Units Other Than Participants: Images
Groups:
- Lateral Image Alone: Lateral x-ray of surgical field viewed alone
- Anteroposterior Image Alone: Anteroposterior x-ray of surgical field viewed alone
- Lateral and Anteroposterior Images Together: Lateral and Anteroposterior x-rays of surgical field view together
Arm/Group | Lateral Image Alone | Anteroposterior Image Alone | Lateral and Anteroposterior Images Together
Number analyzed (Participants) | 111 | 111 | 111
Number analyzed (Images) | 111 | 111 | 111
Cohen's Kappa | 0.76 | 0.73 | 0.80

2. Primary Outcome: Interobserver Reproducibility
Description: Interobserver Reproducibility is the agreement (Cohen's Kappa) between observers interpretations
Time Frame: Intraoperative
Measure: Number; unit: Cohen's Kappa
Units Other Than Participants: Images
Groups:
- Lateral and Anteroposterior Images Together: Lateral and Anteroposterior x-rays of surgical field viewed together
Arm/Group | Lateral Image Alone | Anteroposterior Image Alone | Lateral and Anteroposterior Images Together
Number analyzed (Participants) | 111 | 111 | 111
Number analyzed (Images) | 111 | 111 | 111
Cohen's Kappa | 0.89 | 0.85 | 0.96

3. Primary Outcome: Intraobserver Reproducibility
Description: Intraobserver Reproducibility is the agreement (Cohen's Kapp) of an observer with himself
Time Frame: Intraoperative
Measure: Number; unit: Cohen's Kappa
Units Other Than Participants: Images
Arm/Group | Lateral Image Alone | Anteroposterior Image Alone | Lateral and Anteroposterior Images Together
Number analyzed (Participants) | 111 | 111 | 111
Number analyzed (Images) | 111 | 111 | 111
Cohen's Kappa | 0.91 | 0.88 | 0.96

4. Primary Outcome: Sensitivity
Description: Sensitivity is the percentage of all images appearing to have a sponge in which a sponge was truly present
Time Frame: Intraoperative
Measure: Number; unit: percentage of correct interpretations
Units Other Than Participants: Images
Arm/Group | Lateral Image Alone | Anteroposterior Image Alone | Lateral and Anteroposterior Images Together
Number analyzed (Participants) | 111 | 111 | 111
Number analyzed (Images) | 111 | 111 | 111
percentage of correct interpretations | 82 | 86 | 87

5. Primary Outcome: Specificity
Description: Specificity is the percentage of all images appearing to not have a sponge in which a sponge was truly not present
Time Frame: Intraoperative
Measure: Number; unit: percentage of correct interpretations
Units Other Than Participants: Images
Arm/Group | Lateral Image Alone | Anteroposterior Image Alone | Lateral and Anteroposterior Images Together
Number analyzed (Participants) | 111 | 111 | 111
Number analyzed (Images) | 111 | 111 | 111
percentage of correct interpretations | 95 | 88 | 93

ADVERSE EVENTS:
Time Frame: Intraoperative
Arm/Group | Retained Sponge Group | No Retained Sponge Group
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55
Other Adverse Events (participants affected / at risk) | 0/56 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT04097678/Prot_SAP_000.pdf